CLINICAL TRIAL: NCT02751203
Title: Make Safe Happen App Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lara McKenzie (Other)
Responsible Party: Sponsor-Investigator, Lara McKenzie, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB16-00119
Record Dates: First submitted 2016-03-28; First posted 2016-04-26 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Health Knowledge,Practices,Attitudes

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Make Safe Happen App Intervention (Experimental): Pre- and post-test delivered to online survey panel participants. Instruction to download and use the intervention (Make Safe Happen Mobile App) for 1 week.
  Interventions: Behavioral: Make Safe Happen App
- Make Safe Happen App Control (No Intervention): A subset of online survey panel participants (n=200) will complete a pre- and post-test survey but will receive a non-safety app (e.g. a free recipe app). After the study, participants will be asked to download the intervention app.

INTERVENTIONS:
Behavioral: Make Safe Happen App — The Make Safe Happen app is a mobile app (available for free download android and iOS) developed by the safety experts in the Center for Injury Research and Policy. Parents and caregivers can use the app to learn how to make their homes safer with room-to-room safety checklists and links to recommended products. App users can also create to-do lists, set reminders and track their progress.
  Arms: Make Safe Happen App Intervention

SUMMARY:
Unintentional injury is the leading cause of death for young children in the United States (U.S.) and is responsible for more child deaths than they next three causes combined, that is, homicide, suicide, and cancer. Each year approximately 9,000 children die, 250,000 are hospitalized and more than 9,000,000 children are treated in emergency departments for preventable injuries. Child and adolescent unintentional injury deaths have not declined to the same extent that other diseases have, and resources directed at reducing child injury are not commensurate with the burden it poses. More than 50% of these injuries occur in and around the home, where young children spend most of their time.

Unlike diseases such as cancer, there is no need to wait on a cure...there already is one. Many of these injuries can be prevented through the use of safety equipment and by following safety recommendations. Using known, effective countermeasures can prevent or reduce the consequences of a child being injured yet these devices are not routinely utilized. Barriers related to identifying hazards, finding credible information and recommendations, and obtaining the safety products best-suited to the features of your home make creating a safe home challenging for caregivers. Interventions for increasing home safety behaviors have ranged from educational materials, health care provider counseling, safety product distribution, hands-on experiential learning in a safety resource center--these have all been evaluated with varying degrees of effectiveness, however, wide-reaching interventions to reach large/substantial caregiver audiences, are needed. Offering tailored safety information on multiple topics via a single platform, combined with the ability to acquire safety devices, is a more efficient means to reach a large segment of the population and may help reduce the aforementioned barriers.

Thus, there is an urgent need for mobile technologies to reduce barriers by helping parents identify injury hazards in their homes, consolidate credible injury prevention recommendations, organize information by room or feature, tailor by child age, facilitate the acquisition and installation of safety products, encourage and track progress, thereby increasing the likelihood that parents accomplish these important life-saving safety tasks.

DETAILED DESCRIPTION:
Unintentional injury is the leading cause of death for young children in the United States (U.S.) and is responsible for more child deaths than the next three causes combined, that is, homicide, suicide and cancer. Each year approximately 9,000 children die, 250,000 are hospitalized and more than 9,000,000 children are treated in emergency departments for preventable injuries (at a cost of around $87 billion in medical and societal costs). Child and adolescent unintentional injury deaths have not declined to the same extent as other diseases have, and resources directed at reducing child injury are not commensurate with the burden it poses. More than 50% of these injuries occur in and around the home, where young children spend most of their time. Common causes of fatal and non-fatal unintentional childhood injuries include: fires and burns, falls, drowning, poisoning, and suffocation. For example, residential fires account for nearly 90 percent of all fire-related deaths. Almost 13,000 children are injured by TV tip-overs each year. Medications are the leading causes of child poisoning. Finally, other home hazards include bunk beds, high chairs, windows, stoves and ovens, button batteries, laundry packets, and toys-ubiquitous products and home features present in nearly every U.S. home.

Unlike diseases such as cancer, there is no need to wait on a cure...there already is one. Many of the injuries can be prevented through the use of safety equipment and by following safety recommendations. Using known, effective countermeasures, namely, smoke alarms, carbon monoxide detectors, stair gates, cabinet locks and latches, and anchoring TV and furniture can prevent or reduce the consequences of a child being injured. Unfortunately, overall the rates for these safety behaviors vary/are low (add a citation). Barriers related to identifying hazards, finding credible information and recommendations, and obtaining the safety products best-suited to the features of a home make creating a safe home difficult for parents and caregivers. Interventions for increasing home safety behaviors have ranged from the provision of educational materials, to health care provider counseling, safety product distribution, hands-on experiential learning provided in safety resource centers have been evaluated (with varying degrees of effectiveness), however, wide-reaching interventions, to reach large/substantial parent and caregiver audiences, are needed. Offering tailored safety information on multiple topics via a single platform, combined with the ability to acquire safety devices, is a more efficient means to reach a large segment of the population and may help reduce the aforementioned barriers.

Thus there is an urgent need for mobile technologies-that is, programs using mobile phone or tablet, including apps and text messaging, or portable devices to deliver an intervention-to reduce barriers by helping parents identify injury hazards in their homes, consolidate credible injury prevention recommendations, organize information by room or feature, tailor by child age, facilitate the acquisition and installation of safety products, encourage and track progress, thereby increasing the likelihood that parents accomplish these important and life-saving safety tasks. Our long-term goal is to prevent or reduce the consequences of home-related child injuries. The overall objective of this proposed research, which is the next step toward attainment of our long-term goal, is to preliminarily evaluate a mobile technology-based health behavior change intervention, the Make Safe Happen® app, for improving knowledge and behavior for the prevention of unintentional child injuries. Our central hypothesis is that parents will have increased safety knowledge and more safety behaviors (self-reported and observed), and higher behavioral intention to make their homes safer after utilizing the Make Safe Happen® app compared to a control group. The rationale that underlies the proposed research is derived from the Health Belief Model (HBM) which explains that an individual's perceptions of a threat posed by a health problem (susceptibility, severity), the benefits of avoiding the threat (perceived benefits), and factors influencing the decision to act (barriers, cues to action, and self-efficacy) effect their decision about whether to take action to avoid injury or illness (National Cancer Institute 2005). The investigators plan to objectively test our central hypothesis and, thereby, attain the objective of this application by pursuing the following specific aims:

Specific Aim 1. Determine whether a mobile technology-based health behavior change intervention, the Make Safe Happen® app is effective in improving safety knowledge for the prevention of unintentional child home-related injuries, compared with no intervention. Our working hypothesis is that parents and caregivers receiving the intervention will have greater safety knowledge than parents and caregivers in the control group.

Specific Aim 2. Determine whether a mobile technology-based health behavior change intervention, the Make Safe Happen® app is effective in increasing behavioral intention for the prevention of unintentional child home-related injuries, compared with no intervention or alternate interventions. Our working hypothesis is that parents and caregivers reporting higher behavioral intention will be more likely to complete tasks related to "childproofing" or "safety proofing" their homes.

Specific Aim 3. Preliminarily investigate whether a mobile technology-based health behavior change intervention, the Make Safe Happen® app is effective in improving safety behaviors, acquisition and use of safety devices for the prevention of unintentional child home-related injuries, compared with no intervention.

Possible Exploratory Sub-Aims Sub-aim #1. Evaluate race and ethnicity as a potentially important modifier of the impact of the intervention.

Sub-aim #2: Evaluate household income as a potentially important modifier of the impact of the intervention.

Sub-aim #3: notifications [NOTE: if app use period is only 1 week long, they will not naturally receive notifications as they are currently proposed] Sub-aim #4: e-health literacy (defined as the ability to seek, find, understand, and appraise health information from electronic sources and apply the knowledge gained to addressing or solving a health problem)(Norman and Skinner 2006)

It is anticipated that these aims will yield the following expected outcomes. First, the investigators expect to determine the effect of the intervention on parents' safety knowledge, thereby demonstrating the utility of a mobile app for future unintentional child home-related injury prevention. Second, the investigators expect to learn whether the intervention increases behavioral intention to complete home safety behaviors and safety device acquisition. Third, the investigators will explore whether the intervention increases safety behaviors, acquisition and use of safety devices. In an exploratory aim the investigators will begin to assess whether the intervention is adopted differently among parents of varying races/ethnicities, which will suggest opportunities for tailoring the intervention to maximize its impact. Next, the investigators will have established a link between parents' behavioral intention related to home injury prevention behaviors and device use, which will inform future prevention efforts and expansion of the Make Safe Happen® program and app. Finally, the investigators will provide new insights into the synergism between caring for young children and providing them a safe home environment free of hazards. These outcomes are expected to have an important positive impact because providing a safe home environment has the potential to prevent or reduce unintentional child injuries and deaths, as will now be detailed in the next section.

ELIGIBILITY:
Inclusion Criteria:

* have a smart phone (iOS or Android)
* have willingness to download and install a free mobile application
* parents must be comfortable answering questions online, in English
* parent or legal guardian (male or female) of a child 0-12 years, who lives with them most of the time.

Exclusion Criteria:

* have previously downloaded or used the Make Safe Happen® app.
* have participated in other parts of the study (ie.Online survey participants will not be eligible for participation in the parent focus groups or home observations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5085 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Safety Knowledge Score | 2 weeks
  A safety knowledge score will be calculated by summing the number of correct answers collected from 10-12 questions regarding the participant's safety knowledge. These will be asked at both the pre and post test. Scores will be compared over time and between groups.

SECONDARY OUTCOMES:
Behavioral Intention assessed by using the Health Belief Model | 2 weeks
  A series of questions (10-15) developed with the use of the Health Belief Model will be asked to access the change in behavior intention. Questions will be asked at the pre and post tests and compared over time and between groups.

OTHER OUTCOMES:
Number of safety devices | 2 weeks
  Participants will complete an inventory of the safety devices they have installed or use in their home during the pre and post tests. Number of safety products will be compared over time and between groups.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McKenzie LB, Roberts KJ, McAdams RJ, Abdel-Rasoul M, Kristel O, Szymanski A, Keim SA, Shields WC. Efficacy of a mobile technology-based intervention for increasing parents' safety knowledge and actions: a randomized controlled trial. Inj Epidemiol. 2021 Oct 1;8(1):56. doi: 10.1186/s40621-021-00350-w. PMID 34593040
- [Derived] McKenzie LB, Roberts KJ, Clark R, McAdams R, Abdel-Rasoul M, Klein EG, Keim SA, Kristel O, Szymanski A, Cotton CG, Shields WC. A randomized controlled trial to evaluate the Make Safe Happen(R) app-a mobile technology-based safety behavior change intervention for increasing parents' safety knowledge and actions. Inj Epidemiol. 2018 Mar 12;5(1):5. doi: 10.1186/s40621-018-0133-3. PMID 29527644